CLINICAL TRIAL: NCT04689555
Title: Safety and Efficacy of Femoral Artery Hemostasis Without Manual Compression After Femoral Artery Puncture (FAST): a Prospective, Randomized, Open-label, Controlled, Multicenter Trial
Brief Title: Femoral Artery Hemostasis Without Manual Compression
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Shenghua Zhou, Professor, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAST2020
Record Dates: First submitted 2020-12-24; First posted 2020-12-30 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Femoral Arterial Hemostasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel method without manual compression (Experimental)
  Interventions: Procedure: Novel method without manual compression
- Standard method with manual compression (Active Comparator)
  Interventions: Procedure: Standard method with manual compression.

INTERVENTIONS:
Procedure: Novel method without manual compression — Novel method for femoral artery hemostasis without manual compression. After sheath removal, four or five sterile gauzes were overlaid layer by layer and then bandaged without the procedure of manual compression.
  Arms: Novel method without manual compression
Procedure: Standard method with manual compression. — Standard method for femoral artery hemostasis with manual compression.After sheath removal, manual compression was continued for at least 10 minutes or until hemostasis. After that four or five sterile gauzes were overlaid layer by layer and then bandaged without the procedure of manual compression.
  Arms: Standard method with manual compression

SUMMARY:
FAST trial is a prospective, randomized, controlled, multicenter study in participants needing hemostasis after femoral arterial puncture. All eligible participants will be randomly assigned to either manual compression or novel method without manual compression after femoral arterial puncture. This study is aimed to investigate if novel method without manual compression is noninferior to manual compression regarding access site complications.

DETAILED DESCRIPTION:
The common femoral artery is the most frequently used access site in cardiovascular interventional therapy. Closure of the arteriotomy site is usually achieved by manual compression after femoral arterial puncture. There are many disadvantages of this standard method for hemostasis which is still related to high rate of access-site complications such as pseudoaneurysm, major bleeding, ipsilateral groin hematomas and so on. Several vascular closure devices are emerging as novel means for improving patient comfort and accelerating ambulation after invasive cardiovascular procedures performed via femoral arterial access, however, the cost performance and other aspects limit its wide application especially in developing countries.

Actually the investigators found a novel method for femoral artery hemostasis without manual compression. After sheath removal, four or five sterile gauzes were overlaid layer by layer and then bandaged without the procedure of manual compression.

FAST trial is aimed to investigate if the safety and efficacy of this novel method without manual compression is noninferior to the standard manual compression.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing femoral access cardiovascular interventional therapy
* Patient must be competent for providing informed written consent

Exclusion Criteria:

* Peripheral arterial occlusive disease
* Prior peripheral artery surgery
* Critical limb ischemic
* Femoral arterial intubation failure
* Uncontrolled hypertension >220/110 mmHg
* Coagulopathy (bleeding disorder)
* Local infection
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Composite of arterial access related complications | 1 month
  Composite of arterial access related complications, defined as the composite of:
  * Rate of ipsilateral groin hematomas with largest diameter exceeding 5 cm
  * Pseudoaneurysm
  * AV-Fistula
  * Major bleeding
  * Critical limb ischemia
  * Local infection
  * Need for vascular surgical or interventional treatment

SECONDARY OUTCOMES:
Time to hemostasis | 1 month
  From sheath removal to complete hemostasis
Repeat manual compression | 1 month
  Need for repeated manual compression after end of closure procedure
Total procedure time | 1 month
  From sheath removal to the end of the whole procedure

CONTACTS AND LOCATIONS:
Overall Officials: Shenghua Zhou, Ph.D, Study Chair — Second Xiangya Hospital
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No